CLINICAL TRIAL: NCT03974451
Title: Visual Performance After Trifocal vs Extended Range of Vision Presbyopia-correcting Intraocular Lenses
Brief Title: A Comparison of FineVision Intraocular Lenses vs Symfony Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Finevision vs Symfony IOL
Record Dates: First submitted 2019-04-11; First posted 2019-06-05 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Cataract; Lens Opacities; Presbyopia
Keywords: Intraocular Lens; trifocal; extended range of vision; diffractive achromatic technology
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL implantation experimental (Experimental): Implantation of the PhysIOL FineVision POD F® IOL
  Interventions: Device: IOL implantation experimental
- IOL implantation active comparator (Active Comparator): Implantation of the Abbott Medical Optics, Inc. Tecnis Symfony® IOL.
  Interventions: Device: IOL implantation active comparator

INTERVENTIONS:
Device: IOL implantation experimental — Implantation of of PhysIOL trifocal FineVision® POD F IOL
  Arms: IOL implantation experimental
Device: IOL implantation active comparator — Implantation of the Abbott Medical Optics, Inc. Tecnis Symfony® IOL
  Arms: IOL implantation active comparator

SUMMARY:
This is a prospective randomised open-label study with the aim to compare the visual performance of the trifocal FineVision® IOL versus the extended range of vision Symfony® IOL after phaco-emulsification cataract surgery.

DETAILED DESCRIPTION:
With the advent of a new intraocular lens (IOL) materials, technologies and advanced optics, higher spectacle independence after surgery is now possible.

Multifocal IOLs work by splitting light into different foci, which is known to generate photic effects. Trifocal optics, which have been available on the European market since 2010, offer spectacle independence in most cases. Typically, visual acuity is maintained throughout the whole range of vision from distance to near vision, and general patient satisfaction has proven that trifocal IOLs are well tolerated by patients.

Patients having irregular corneal astigmatism, large pupils and weak zonules were considered unsuitable candidates for multifocal IOLs, while patients who aim for spectacle independence and with low pre-operative regular astigmatism were considered to be good candidates.

The Fine Vision IOL (PhysIOL®; Liège, Belgium) is a diffractive trifocal IOL that provides an intermediate focus at 1.75 D and a near focus at 3.5 D (both at the IOL plane). This corresponds to a nominal intermediate add of approximately +1,15 D and near add of about 2,25 D at the corneal plane, depending on the geometry of the patient's eye. This intermediate focal point is expected to improve patient satisfaction relative to bifocal IOLs, since bifocal IOLs have a greater drop off in visual acuity (VA) in the intermediate range. There is a concern that the addition of a third focal point may increase halos, However, a relatively small percentage of energy is dedicated to intermediate vision when compared to distance and near vision. The trifocal diffractive structure asymmetrically directs incident light to distant (50%) intermediate (20%) and near (30%) focal points, independent of pupil diameter (up to 4,5 mm).

The FineVision is an aspheric trifocal IOL composed of 25% hydrophilic acrylic material with a blue light and ultraviolet light blocker. It has a total diameter of 10,75 mm and an optic body diameter of 6,15 mm.

The Tecnis Symfony is an extended range of vision IOL based on diffractive achromatic technology. The IOL has an achromatic diffractive pattern that elongates the focus and compensates for the chromatic aberration of the cornea. According to the manufacturer, halos are not expected with this IOL, because it provides an elongated focal area rather than one or various focal points. The IOL has a biconvex wavefront-designed anterior aspheric surface and a posterior achromatic diffractive surface. The total diameter of the IOL is 13.0 mm, and the optic zone diameter is 6.0 mm. It is an ultraviolet-filtering hydrophobic acrylic material with a refractive index of 1,47 at 35° C.

This is a prospective randomised open-label study with the aim to compare the visual performance of the trifocal FineVision® IOL versus the extended range of vision Symphony® IOL after phaco-emulsification cataract surgery.

All patients will undergo and complete preoperative ophthalmologic examinations including refractive status, uncorrected and corrected near and distance visual acuities, biometry and keratometry.

Postoperative, all patients will receive topical antibiotic treatment for 1 week and topical steroid tapered treatment for 4 weeks as well as NSAID topical treatment for 4 weeks. All patients will be followed up after 2 days, 1 week and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Cataract patients requesting independence from spectacles
2. Potential visual acuity of 0.0 logMar

Exclusion Criteria:

1. Unrealistic expectations (sharp clear vision is the main concern of the patient)
2. Ocular pathology besides cataract (glaucoma, macular degeneration, retinopathies, corneal opacities, corneal guttata.. etc.)
3. Previous refractive surgery
4. Expected pathology after surgery (p.e. uveitis, diabetic retinopathy, PEX)
5. Preoperative corneal astigmatism of > 1.0 D
6. Any intraocular or postoperative complication
7. Dry eye disease
8. History of ocular trauma

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Corrected Distance Visual Acuity at 6m (CDVA) - monocular | 3 months postoperative
  CDVA is measured with ETDRS charts placed in 6m distance with best aided corrective glasses according to International Standards Organization (ISO) 11979-7:2014. This assessment is done monocularly.

SECONDARY OUTCOMES:
Uncorrected Distance Visual Acuity at 6m (UDVA) - monocular | 3 months postoperative
  UDVA is measured with ETDRS charts placed in 6m distance according to International Standards Organization (ISO) 11979-7:2014. This assessment is done monocularly.
Uncorrected Intermediate Visual Acuity at 65cm (UIVA) - monocular | 3 months postoperative
  UIVA is measured with ETDRS charts placed in 65cm distance. The examination is done without corrective glasses and according to International Standards Organization (ISO) 11979-7:2014. This assessment is done monocularly.
Distance Corrected Intermediate Visual Acuity at 65cm (DCIVA) - monocular | 3 months postoperative
  DCIVA is measured with ETDRS charts placed in 65cm distance with corrective glasses for far distance according to International Standards Organization (ISO) 11979-7:2014. This assessment is done monocularly.
Uncorrected Near Visual Acuity at 35cm (UNVA) | 3 months postoperative
  UNVA is measured with ETDRS charts placed in 35cm distance. The examination is done without corrective glasses and according to International Standards Organization (ISO) 11979-7:2014. This assessment is done monocularly.
Distance Corrected Near Visual Acuity at 35cm (DCNVA) - monocular | 3 months postoperative
  DCNVA is measured with ETDRS charts placed in 35cm distance with corrective glasses for far distance according to International Standards Organization (ISO) 11979-7:2014. This assessment is done monocularly.
Defocus Curve | 3 months postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -4.0 D to 0.0 D. This examination is performed monocularly.
Contrast Sensitivity | 3 months postoperative
  Contrast Sensitivity under photopic light conditions using the CSV-1000 contrast test.
National Eye Institute Visual Functioning Questionnaire - 25 (VFQ-25) | 3 months postoperative
  For this study, the validated and verified questionnaire VFQ-25 (National Eye Institute) will be used. The VFQ-25 consists of a base set of 25 vision- targeted questions representing 11 vision-related constructs (General Health, General Vision, Ocular Pain,Near Activities, Distance Activities, Vision Specific (Social Functioning, Mental Health, Role Difficulties, Dependency), Driving, Color Vision, Peripheral Vision), plus an additional single-item general health rating question.
  The minimum score is 0 and the maximum score is 100 for each construct. Higher values represent a better outcome.
Manifest Refraction | 3 months postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to International Standards Organization (ISO) 11979-7:2014.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed H. F. Ghoneem, MD, Principal Investigator — Department of Ophthalmology, Faculty of Medicine, University of Alexandria,
Locations (1):
- Department of Ophtalmology, Alexandria Main University Hospital (AMUH), Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No